CLINICAL TRIAL: NCT00577720
Title: Study to Assess the Efficacy, Safety and Pharmacokinetics of Risedronate Upon Oral Administration of a 35 mg Delayed-Release, a 50 mg Delayed-Release or a 35 mg Immediate-Release Administered Weekly for 13 Weeks to Postmenopausal Women
Brief Title: Assess the Safety, Efficacy, and Pharmacokinetics of Immediate and Delayed Release Weekly Risedronate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005107
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Results first posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2011-11

CONDITIONS: Postmenopausal Women
MeSH Terms: interventions — Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 35 mg IRBB (Active Comparator): 35 mg immediate release risedronate tablet, 30 minutes prior to breakfast, once a week for 13 weeks
  Interventions: Drug: risedronate
- 35 mg DRFB (Experimental): 35 mg delayed release risedronate tablet, immediately following breakfast, once a week for 13 weeks
  Interventions: Drug: risedronate
- 50 mg DRFB (Experimental): 50 mg delayed release risedronate tablet, immediately following breakfast, once a week for 13 weeks
  Interventions: Drug: risedronate
- 50 mg DRBB (Experimental): 50 mg delayed release risedronate tablet, 30 minutes prior to breakfast, once a week for 13 weeks
  Interventions: Drug: risedronate

INTERVENTIONS:
Drug: risedronate — 35mg immediate release risedronate tablet before breakfast, once a week for 13 weeks
  Arms: 35 mg IRBB
Drug: risedronate — 35mg delayed release risedronate tablet following breakfast, once a week for 13 weeks
  Arms: 35 mg DRFB
Drug: risedronate — 50mg delayed release risedronate tablet following breakfast, once a week for 13 weeks
  Arms: 50 mg DRFB
Drug: risedronate — 50mg delayed release risedronate tablet before breakfast, once a week for 13 weeks
  Arms: 50 mg DRBB

SUMMARY:
To compare the efficacy 50 mg delayed-release risedronate tablet, dosed immediately after breakfast, to a 35 mg immediate-release tablet, administered according to labeling instructions.

DETAILED DESCRIPTION:
To compare the efficacy, based on the bone turnover marker (BTM) serum Type I collagen C-telopeptide (CTx), of a 50 mg delayed-release risedronate tablet, administered immediately after a typical breakfast, to that of a 35 mg immediate-release tablet, administered according to labeling instructions (ie, at least 30 minutes prior to breakfast) in postmenopausal women after 13 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* In generally good health, as determined by medical history, physical examination, and laboratory test results
* Postmenopausal greater than 2 years, naturally or surgically based on medical history.

Exclusion Criteria:

* Used any of the following medications within 3 months prior to dosing or used any of the following medications for more than 1 month at any time within 6 months prior to dosing:

  * oral or parenteral glucocorticoids (5 mg prednisone or equivalent/day)
  * anabolic steroids
  * estrogens (oral, skin patch, or gel), except for low dose vaginal products or insertable estrogen ring, selective estrogen-receptor modulators, or estrogen-related drugs
  * progestins
  * calcitonin
  * vitamin D supplements
  * calcitriol, calcidiol, or alfacalcidol at any dose
  * any bisphosphonate
  * fluoride
  * strontium
  * parathyroid hormone, including teriparatide

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2006-07; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lu A Sun, MD, PhD, Study Director — Procter and Gamble
Locations (6):
- United States (6):
  - Research Facility, Costa Mesa, California
  - Research Facility, Gainsville, Florida
  - Research Facility, Miami, Florida
  - Research Facility, Honolulu, Hawaii
  - Research Site, Dallas, Texas
  - Research Facility, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Screening began 14-Jul-2006
Groups:
- 35 mg IRBB (Immediate Release Before Breakfast): 35 mg immediate release risedronate tablet, 30 minutes prior to breakfast, once a week for 13 weeks
- 35 mg DRFB (Delayed Release Following Breakfast): 35 mg delayed release risedronate tablet, immediately following breakfast, once a week for 13 weeks
- 50 mg DRBB (Delayed Release Before Breakfast): 50 mg delayed release risedronate tablet, 30 minutes prior to breakfast, once a week for 13 weeks
Period: Overall Study
Arm/Group | 35 mg IRBB (Immediate Release Before Breakfast) | 35 mg DRFB (Delayed Release Following Breakfast) | 50 mg DRFB | 50 mg DRBB (Delayed Release Before Breakfast)
Started | 37 | 36 | 36 | 72
ITT (Intent to Treat) Population | 34 | 35 | 35 | 65
Completed | 33 | 35 | 35 | 65
Not Completed | 4 | 1 | 1 | 7
Not completed — Adverse Event | 2 | 1 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 35 mg IRBB (Immediate Release Before Breakfast) | 35 mg DRFB (Delayed Release Following Breakfast) | 50 mg DRFB | 50 mg DRBB (Delayed Release Before Breakfast) | Total
Number analyzed (Participants) | 37 | 36 | 36 | 72 | 181
Age Continuous [Mean (Standard Deviation); unit: years] | 61.1 (6.2) | 58.9 (6.7) | 60.0 (6.1) | 59.7 (7.8) | 59.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 36 | 72 | 181
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 14 | 23 | 59
  Not Hispanic or Latino | 24 | 27 | 22 | 49 | 122
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (Oriental) | 6 | 6 | 3 | 10 | 25
  Black | 0 | 1 | 3 | 2 | 6
  Caucasian | 30 | 29 | 26 | 56 | 141
  Multi-Racial | 0 | 0 | 0 | 1 | 1
  Other | 1 | 0 | 4 | 2 | 7
  Hawaiian/Pacific Islander | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 37 | 36 | 36 | 72 | 181

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Serum CTX (Type I Collagen C-telopeptide), ITT (Intent to Treat) Population
Time Frame: Baseline and Week 13
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 35 mg IRBB (Immediate Release Before Breakfast) | 35 mg DRFB (Delayed Release Following Breakfast) | 50 mg DRFB | 50 mg DRBB (Delayed Release Before Breakfast)
Number analyzed (Participants) | 34 | 35 | 35 | 65
Percent Change | -43.20 [-55.83 to -30.58] | -62.08 [-73.59 to -50.56] | -65.11 [-77.70 to -52.52] | -66.30 [-77.42 to -55.18]
Statistical Analysis 1: Comparison: 35 mg IRBB (Immediate Release Before Breakfast) vs 35 mg DRFB (Delayed Release Following Breakfast); For power calculations, assumed that variability in test treatment groups is no more than 50% higher than reference group. If true ratio of CTX is 0.65, the power to detect this departure from a ratio of 1.0 in the primary analysis is 0.88; Test type: Superiority or Other; Ratio (LS Mean 35 mg DRFB/35 mg IRBB) = 1.437, 90% CI 2-sided [1.091 to 1.964]
Statistical Analysis 2: Comparison: 35 mg IRBB (Immediate Release Before Breakfast) vs 50 mg DRBB (Delayed Release Before Breakfast); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRBB/35 mg IRBB) = 1.507, 90% CI 2-sided [1.139 to 2.066]
Statistical Analysis 3: Comparison: 35 mg IRBB (Immediate Release Before Breakfast) vs 50 mg DRFB; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRFB/35 mg IRBB) = 1.535, 90% CI 2-sided [1.177 to 2.086]
Statistical Analysis 4: Comparison: 35 mg DRFB (Delayed Release Following Breakfast) vs 50 mg DRFB; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRFB/50 mg DRBB) = 1.068, 90% CI 2-sided [0.867 to 1.321]
Statistical Analysis 5: Comparison: 50 mg DRFB vs 50 mg DRBB (Delayed Release Before Breakfast); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRFB/50 mg DRBB) = 1.018, 90% CI 2-sided [0.824 to 1.267]

2. Secondary Outcome: Percent Change in Urine NTX/Cr (Urine Type I Collagen Cross-linked N-telopeptide Corrected for Creatinine Clearance), ITT Population
Time Frame: Baseline and Week 13
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 35 mg IRBB (Immediate Release Before Breakfast) | 35 mg DRFB (Delayed Release Following Breakfast) | 50 mg DRFB | 50 mg DRBB (Delayed Release Before Breakfast)
Number analyzed (Participants) | 34 | 35 | 35 | 65
Percent Change | -38.57 [-56.60 to -20.54] | -46.60 [-63.04 to -30.17] | -43.65 [-61.62 to -25.67] | -54.27 [-70.14 to -38.40]
Statistical Analysis 1: Comparison: 35 mg IRBB (Immediate Release Before Breakfast) vs 35 mg DRFB (Delayed Release Following Breakfast); The target numbers of subjects assessable for the primary analysis are 70 in the 50 mg DRFB group and 35 in the 35 mg IRBB group. Sample sizes are determined to provide adequate power for the primary comparison (ie, serum CTX for 50 mg DRFB vs. 35 mg IRBB); Test type: Superiority or Other; Ratio (LS Mean 35 mg DRFB/35 mg IRBB) = 1.208, 90% CI 2-sided [0.749 to 2.099]
Statistical Analysis 2: Comparison: 35 mg IRBB (Immediate Release Before Breakfast) vs 50 mg DRBB (Delayed Release Before Breakfast); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRBB/35 mg IRBB) = 1.132, 90% CI 2-sided [0.665 to 2.003]
Statistical Analysis 3: Comparison: 35 mg IRBB (Immediate Release Before Breakfast) vs 50 mg DRFB; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRFB/35 mg IRBB) = 1.407, 90% CI 2-sided [0.913 to 2.404]
Statistical Analysis 4: Comparison: 35 mg DRFB (Delayed Release Following Breakfast) vs 50 mg DRFB; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRFB/35 mg DRFB) = 1.165, 90% CI 2-sided [0.797 to 1.752]
Statistical Analysis 5: Comparison: 50 mg DRFB vs 50 mg DRBB (Delayed Release Before Breakfast); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRFB/50 mg DRBB) = 1.243, 90% CI 2-sided [0.828 to 1.990]

3. Secondary Outcome: Percent Change in Serum BAP (Bone-specific Alkaline Phosphatase), ITT Population
Time Frame: Baseline and Week 13
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | 35 mg IRBB (Immediate Release Before Breakfast) | 35 mg DRFB (Delayed Release Following Breakfast) | 50 mg DRFB | 50 mg DRBB (Delayed Release Before Breakfast)
Number analyzed (Participants) | 34 | 35 | 35 | 65
Percent Change | -10.99 [-19.62 to -2.365] | -10.41 [-18.28 to -2.545] | -20.00 [-28.60 to -11.40] | -17.36 [-24.96 to -9.767]
Statistical Analysis 1: Comparison: 35 mg IRBB (Immediate Release Before Breakfast) vs 35 mg DRFB (Delayed Release Following Breakfast); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 35 mg DRFB/35 mg IRBB) = 0.947, 90% CI 2-sided [0.316 to 2.993]
Statistical Analysis 2: Comparison: 35 mg IRBB (Immediate Release Before Breakfast) vs 50 mg DRBB (Delayed Release Before Breakfast); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRBB/35 mg IRBB) = 1.820, 90% CI 2-sided [0.929 to 5.429]
Statistical Analysis 3: Comparison: 35 mg IRBB (Immediate Release Before Breakfast) vs 50 mg DRFB; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRFB/35 mg IRBB) = 1.580, 90% CI 2-sided [0.801 to 4.718]
Statistical Analysis 4: Comparison: 35 mg DRFB (Delayed Release Following Breakfast) vs 50 mg DRFB; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRFB/35 mg DRFB) = 1.668, 90% CI 2-sided [0.856 to 4.668]
Statistical Analysis 5: Comparison: 50 mg DRFB vs 50 mg DRBB (Delayed Release Before Breakfast); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Ratio (LS Mean 50 mg DRFB/50 mgDRBB) = 0.868, 90% CI 2-sided [0.504 to 1.488]

ADVERSE EVENTS:
Time Frame: 14 Jul 2006 thru 27 Jan 2007
Arm/Group | 35 mg IRBB (Immediate Release Before Breakfast) | 35 mg DRFB (Delayed Release Following Breakfast) | 50 mg DRFB | 50 mg DRBB (Delayed Release Before Breakfast)
Serious Adverse Events (participants affected / at risk) | 0/37 | 1/36 | 0/36 | 1/72
Other Adverse Events (participants affected / at risk) | 27/37 | 19/36 | 24/36 | 51/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 35 mg IRBB (Immediate Release Before Breakfast) (N=37) | 35 mg DRFB (Delayed Release Following Breakfast) (N=36) | 50 mg DRFB (N=36) | 50 mg DRBB (Delayed Release Before Breakfast) (N=72)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 35 mg IRBB (Immediate Release Before Breakfast) (N=37) | 35 mg DRFB (Delayed Release Following Breakfast) (N=36) | 50 mg DRFB (N=36) | 50 mg DRBB (Delayed Release Before Breakfast) (N=72)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 0 (0) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 5 (7)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2) | 1 (1) | 2 (2)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 8 (11)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (4) | 6 (9)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 2 (3) | 0 (0) | 4 (4)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (2) | 4 (4) | 9 (13)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 6 (6) | 7 (14)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (5)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Rectal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 7 (9) | 8 (11) | 10 (10) | 16 (26)
Sinus Headache (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (10)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Herpes Zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes Simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (3)
Gingival Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Cholesterol Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Sodium Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Triglycerides Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less